CLINICAL TRIAL: NCT05530915
Title: Guayusa: The Effect of an Herbal Extract on Alertness and Mental Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2113
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Attention Difficulties
Keywords: mental fatigue; alertness; cognitive; COMPASS; guayusa; energy; fatigue; mood; memory
MeSH Terms: conditions — Mental Fatigue; Fatigue | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active capsule 1: Lower dose guayusa ingredient (Experimental): Oral administration of 175 mg guayusa extract providing 35 mg caffeine
  Interventions: Other: Gel capsule
- Active capsule 2: Higher dose guayusa ingredient (Experimental): Oral administration of 300 mg guayusa extract providing 60 mg caffeine
  Interventions: Other: Gel capsule
- Placebo capsule (Placebo Comparator): Oral administration of 0 mg guayusa extract, 0 mg caffeine. Capsule color-matched to actives 1 and 2 to disguise potential differences in color of contents.
  Interventions: Other: Gel capsule

INTERVENTIONS:
Other: Gel capsule — Single capsule per dose

SUMMARY:
The primary objective of this randomized, double-blind, placebo-controlled, cross-over study is to assess the acute effects of a novel ingredient, guayusa on alertness and mental fatigue compared to a placebo. This trial will utilize the COMPASS cognitive task and cognitive demand battery (CDB) and mood, motivation, and energy measures with assessments taking place at baseline, 60- and 120-minutes post treatment on three separate testing days separated by ~7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-55 years of age, inclusive at Visit 1 (Day -7).
2. BMI <30 kg/m2 at Visit 1 (Day -7).
3. Self-reported poor attention during pre-screening phone call prior to Visit 1 (Day -7).
4. Willing to abstain from alcohol and vigorous physical activity 24 h prior to Visits 1, 2, 3, and 4 (Days -7, 0, 7, and 14).
5. Willing to abstain from all exercise the morning of Visits 1, 2, 3, and 4 (Days -7, 0, 7, and 14).
6. Willing and able to comfortably abstain from caffeine for 24 h prior to Visits 1, 2, 3, and 4 (Days -7, 0, 7, and 14).
7. Non-user of nicotine products (e.g., cigarettes, patches/gum, etc.) within 60 days of Visit 1 (Day-7).
8. Non-user of marijuana and hemp products including CBD products within 60 days of Visit 1 (Day-7).
9. Willing to abstain from over-the-counter drugs or supplements that have stimulating (e.g., containing caffeine or guayusa), cognition boosting, or sedating (e.g., sleeping aids, anti-histamines, decongestants) effects (Appendix 1) for 24 h prior to and during all visits.
10. Willing to maintain habitual diet (including fluids, caffeine, and alcohol), physical activity patterns, sleeping patterns (3 days before each test visit), and body weight throughout the trial.
11. Willing to maintain habitual intake of approved vitamins and supplements throughout the study except during Visits 2, 3, and 4 (Days 0, 7, and 14) whereby participants are required to abstain from any supplements until the end of the study visits.
12. Has no health conditions that would prevent him or her from fulfilling the study requirements or affect study outcomes as judged by the Principal Investigator on the basis of medical history and routine laboratory test results.
13. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Principal Investigator.

Exclusion Criteria:

1. Unable to understand and/or completely perform the practice test to standard minimum requirements and based on queries performed following the practice test at Visit 1 (Day -7).
2. Visual impairments that cannot be corrected with glasses or contact lenses.
3. Known intolerance, allergy, or sensitivity to caffeine or any of the other ingredients in the study products and/or any ingredients of the standardized snack provided, including shellfish, egg, fish, gluten, milk, peanuts, soy, tree nuts (coconut and walnut), and gelatin.
4. Extreme dietary habits (e.g., intermittent fasting, low carbohydrate diet) that would affect study outcomes as judged by the Principal Investigator.
5. Unstable dose of prescription medications (stable is defined as same dose for the past 90 d prior to Visit 1; Day -7).
6. Use of prescription drugs (stable or unstable) that have stimulating (e.g., amphetamines [Adderall® and Dexedrine®], methylphenidate [Concerta® and Ritalin®], diet aids [such as Didrex®, Bontril®, Preludin®, Fastin®, Adipex P®, Ionomin®, and Meridia®], containing caffeine or guayusa), cognition boosting, or sedating (e.g., sleeping aids, drugs to treat mental health disorders) effects.
7. For females on hormone therapy (including oral contraceptives), the subject must be on a stable dose of hormones (defined as same dose for the past 90 d prior to Visit 1; Day -7).
8. Signs or symptoms of an active infection of clinical relevance (e.g., urinary tract or respiratory) within 5 d prior to Visits 2, 3, and 4 (Days 0, 7, and 14). If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved (at the discretion of the Principal Investigator) at least 5 d prior to testing, unless the visit will be out of window. If the visit will be out of window, subjects should continue with testing and a protocol deviation will be required.
9. Experienced evidence of delirium, confusion, or other disturbances of consciousness to the degree that could affect study outcomes, in the judgement of the Principal Investigator.
10. History of learning and/or behavioral disorders such as dyslexia or diagnosed attention deficit hyperactive disorder (ADHD).
11. Neurologic disorder that could produce cognitive deterioration including, but not limited to, Alzheimer's disease, Parkinson's disease, stroke, intracranial hemorrhage, local brain lesions including tumors, and normal pressure hydrocephalus.
12. History of any infective or inflammatory brain disease, including those of viral, fungal, or syphilitic etiologies.
13. History of frequent (≥ 1 occasion/month) migraines that require medication.
14. History of repeated minor head injury (e.g., in boxing) or a single injury resulting in a period of unconsciousness for 1 h or more.
15. History or presence of clinically uncontrolled important endocrine (including hyperparathyroidism, type 1 or 2 diabetes mellitus and/or hypoglycemia), cardiovascular (including, but not limited to history of myocardial infarction, peripheral arterial disease,), pulmonary (including uncontrolled asthma), hepatic, renal, gastrointestinal, hematologic, immunologic, dermatologic, rheumatic (including gout), and/or biliary, that, in the opinion of the Principal Investigator, could interfere with the interpretation of the study results.
16. History or presence of cancer in the prior two years, except for non-melanoma skin cancer.
17. History of major physical trauma (e.g., required hospitalization) or mental trauma (e.g., abuse) within 6 months of Visit 1 (Day -7).
18. Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) as defined by the blood pressure measured at Visit 1 (Day -7). One re-test will be allowed on a separate day prior to Visit 2 (Day 0), for subjects with abnormal blood pressure.
19. Heavy consumer of caffeinated beverages (>400 mg caffeine/d from caffeine-containing products; Appendix 2).
20. Sleep disorder (e.g., sleep apnea) or occupation where sleep during the overnight hours is irregular (e.g., 3rd shift of overnight workers).
21. Female who is pregnant, planning to be pregnant during the study period, or lactating,
22. Female of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation.
23. Exposure to any non-registered drug product or has participated in another intervention study within 30 d prior to Visit 1 (Day -7).
24. Recent history of (within 12 months of screening; Visit 1; Day -7) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
25. Has a condition the Principal Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Mental alertness | Change from pre-dose baseline to 60 minutes post-guayusa consumption compared to placebo
  Current subjective alertness rating on a Visual Analog Scale (VAS) in the COMPASS Cognitive Demand Battery (CDB) by marking on a 100-mm line with the end points labelled "not at all" (left hand end) and "extremely" (right hand end). Scores are calculated as percentage along the line from left to right. Increased alertness is better.

OTHER OUTCOMES:
Mental alertness | Change from pre-dose baseline to 120 minutes post-guayusa consumption compared to placebo.
  Current subjective alertness rating on a Visual Analog Scale (VAS) in the COMPASS Cognitive Demand Battery (CDB) by marking on a 100-mm line with the end points labelled "not at all" (left hand end) and "extremely" (right hand end). Scores are calculated as percentage along the line from left to right. Increased alertness is better.
Mental fatigue | Change from pre-dose baseline to 60 minutes and 120 minutes post-guayusa consumption compared to placebo
  Current subjective alertness rating on a Visual Analog Scale (VAS) in the COMPASS Cognitive Demand Battery (CDB) by marking on a 100-mm line with the end points labelled "not at all" (left hand end) and "extremely" (right hand end). Scores are calculated as percentage along the line from left to right. Decreased mental fatigue is better.
Energy & Fatigue State (EFS) Scales | Change from pre-dose baseline to 60 minutes and 120 minutes post-guayusa consumption compared to placebo
  Rating of current subjective feelings from none to strongest ever felt for physical energy, physical fatigue, mental energy, and mental fatigue. Each EFS-State scale dimension is comprised of answers from three items that are presented and then summed to composite scores ranging from 0 to 300 in the COMPASS Cognitive Demand Battery (CDB). Increased energy and lower fatigue is better.
Mood | Change from pre-dose baseline to 60 minutes and 120 minutes post-guayusa consumption compared to placebo
  Bond-Lader Visual Analog Scale (VAS) in the COMPASS Cognitive Demand Battery, (CDB). 16 scales anchored at either side by an adjective describing a mood, to click at a point on the scale that represents the feeling at that point in time, scored from 0-100. From these 16 scales, three composite scores are calculated describing feelings of 'Alert', 'Calm' and 'Content'. Improved mood is better.
Cognitive test Serial Subtraction | Change from pre-dose baseline to 60 minutes and 120 minutes post-guayusa consumption compared to placebo
  Serial 3s and Serials 7s in the COMPASS Cognitive Demand Battery (CDB). A random starting number (between 800 and 999) is displayed on the screen. Participants are required to subtract a number (e.g. 7s or 3s) from this and continue to subtract from the resultant numbers for the duration of the task. Higher accuracy is better.
Cognitive test RVIP | Change from pre-dose baseline to 60 minutes and 120 minutes post-guayusa consumption compared to placebo
  Rapid Visual Information Processing (RVIP) in the COMPASS Cognitive Demand Battery (CDB). A series of numbers are displayed individually on the screen in quick succession (at a rate of 100 numbers per minute) and participants are required to respond when they see 3 odd numbers in a row or 3 even numbers in a row. Higher accuracy is better.
Cognitive memory test: Words | Change from pre-dose baseline to 60 minutes and 120 minutes post-guayusa consumption compared to placebo
  Accuracy and reaction time for delayed word recall and delayed word recognition in the COMPASS Cognitive Demand Battery (CDB). Higher accuracy and faster reaction time are better.
Cognitive memory test: Pictures | Change from pre-dose baseline to 60 minutes and 120 minutes post-guayusa consumption compared to placebo
  Accuracy and reaction time for delayed picture recognition in the COMPASS Cognitive Demand Battery (CDB). Higher accuracy and faster reaction time is better.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Beckman, MD, Principal Investigator — Mérieux NutriSciences
Locations (1):
- Biofortis Innovation Services, Division of Merieux NutriSciences, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No